CLINICAL TRIAL: NCT02085187
Title: Early Telemedicine Training and Counselling After Hospitalization in Patients With Severe Chronic Obstructive Pulmonary Disease: A Feasibility Study
Brief Title: Early Telemedicine Training in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Lisbeth Rosenbek Minet, Assistent Professor, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-20110036
Record Dates: First submitted 2014-03-06; First posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Pulmonary rehabilitation; Training; Counselling; Telemedicine; Videoconference; COPD; Chronic disease; Internet.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Chronic Disease | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telemedicine training and counselling (Experimental)
  Interventions: Other: Telemedicine training and counselling

INTERVENTIONS:
Other: Telemedicine training and counselling — Training and counselling by the physiotherapist consisted of 3 weekly sessions, lasting 30-45 minutes, over a 3 week period, i.e. a total of 9 supervised sessions. Heart rate and oxygen saturation were monitored during the exercise training. This included thoracic mobilization exercises, cardio training, strength training and breathing exercises. The training intensity was progressed continuously.
  There were 1-2 sessions with the occupational therapist, which consisted of training and counselling on energy conservation techniques. The first session was 60 minutes long and included assessment, counselling and training. This session was delivered in the second week of the intervention. The intervention concluded in the third week, with sessions of 30 minutes as required.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a widespread disease that can have a major impact on the lives of individuals. An essential element in the treatment of COPD is rehabilitation of which supervised training is an important part. However, not all individuals with severe COPD can participate in the rehabilitation provided by hospitals and municipal training centres due to distance to the training venues and transportation difficulties. The aim of the feasibility study was to evaluate an individualised home based training and counselling programme via video conference to patients with severe COPD after hospitalization with regard to safety, clinical outcomes, patients' perception, organisational aspects and economic aspects.

ELIGIBILITY:
Inclusion Criteria:

* severe and very severe COPD (i.e. with an FEV1 (forced expiratory volume in 1 second) value under 50% of the predicted value, an FEV1/FVC (forced vital capacity) ratio < 70%, MRC (Medical Research Council Dyspnoea Scale) grade 3)
* ≥40 years
* hospitalization with exacerbation of COPD
* declined participation in the hospital based rehabilitation
* participation in videoconference sessions with a nurse for one week immediately after discharge.

Exclusion Criteria:

* inability to communicate via telephone and computer
* systolic BP <100mm Hg
* X-rays of the thorax showing abnormalities suspicious of thoracic malignancy or lobar pneumonia
* a diagnosis of cancer or recurrence of cancer within the last 5 years
* hospitalization with septic shock, acute myocardial infarction (AMI) or other serious medical conditions (e.g. kidney disorder)
* heart failure (EF<30%)
* if the patient did not wish to participate.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Clinical COPD Questionnaire (CCQ) | Up to 3 weeks
  A self-administered validated questionnaire measuring the health status of patients with COPD.
Timed Up & Go test (TUG) | Up to 3 weeks
  Measuring the time in seconds (with 2 decimals), it takes a person to rise from an ordinary chair (with back and armrest), walk 3 meters, turn around and walk back to the chair and sit down again
The five time sit to stand test (FTSST) | Up to 3 weeks
  Measures functional lower limb muscle strength, where the time in seconds (2 decimals) used for 5 times rising from a chair is measured.
Patients' falls during training | Up to 3 weeks
Need for acute contact to the general practitioner | Up to 3 weeks
Patient subjective perception | Up to 3 weeks
  The patients submitted a postcard with information about their experience. The postcard was an open ended question and was printed with the text "Dear Department of rehabilitation. My experience of training and counselling by use of the Patient briefcase was … ".
Costs per patient participating in the telemedicine rehabilitation | Up to 3 weeks
  This included renting of the "patient briefcase", establishing of a safe line for data transmission and use of hospital staff.
Reimbursement to the hospital | Up to 3 weeks
  Estimated as the DRG (Diagnose Related Groups) value of the rehabilitation activity similar to the payment for the activity from the regional health system (The Region of Southern Denmark) to the hospital in accordance with health care financing system).
Focus Group interview | Up to 3 weeks
  The perception of the hospital staff of the telemedicine intervention programme was assessed by a focus group interview with the occupational- and physiotherapists who carried out the telemedicine rehabilitation training and thus were familiar with the programme.

CONTACTS AND LOCATIONS:
Overall Officials: Lilian Møllegård, Reg. Nurce, Study Chair — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633
- [Derived] Rosenbek Minet L, Hansen LW, Pedersen CD, Titlestad IL, Christensen JK, Kidholm K, Rayce K, Bowes A, Mollegard L. Early telemedicine training and counselling after hospitalization in patients with severe chronic obstructive pulmonary disease: a feasibility study. BMC Med Inform Decis Mak. 2015 Feb 7;15:3. doi: 10.1186/s12911-014-0124-4. PMID 25886014